CLINICAL TRIAL: NCT04358887
Title: Effect of Piezoelectric Surgery on Quality of Life and Periradicular Healing After Endodontic Surgery : A Randomized Clinical Trial
Brief Title: Effect of Piezoelectric Surgery on Quality of Life and Periradicular Healing After Endodontic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr.Jaya Bharathi
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Periapical Disease
Keywords: piezoelectric surgery, quality of life, hemostasis
MeSH Terms: conditions — Periapical Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- periapical surgery with piezo. (Experimental): After flap reflection bone and root end cutting are done with US6 piezoelectric surgical insert
  Interventions: Procedure: piezoelectric surgery
- Periapical surgery with bur. (Active Comparator): After flap reflection bone and root end cutting are done with surgical bur.
  Interventions: Procedure: conventional bur

INTERVENTIONS:
Procedure: piezoelectric surgery — after flap reflection bone and root end cutting are done with piezoelectric surgical insert
  Arms: periapical surgery with piezo.
Procedure: conventional bur — after flap reflection bone and root end cutting are done with surgical bur
  Arms: Periapical surgery with bur.

SUMMARY:
This study will compare the effect of piezo Vs bur on quality of life and healing after endodontic surgery.

DETAILED DESCRIPTION:
The goal of endodontic surgery has changed from mere reduction of periapical pathosis and preservation of periodontium to successful postoperative management of patient regarding function and esthetics, improving the quality of life of patient and their overall acceptance. Piezoelectric bone surgery is a recent and innovative technology, permitting selective cutting of mineralized tissues sparing soft tissues.In this study after thorough clinical & radiographic examination patients will be given informed consent after explaining the treatment procedure and its associated risks and benefits. Patients are allocated into 2 groups, group 1(piezo group) in which after flap reflection bone cutting and root end cutting are performed with US6 piezoelectric insert and in group 2(control) bone and root end cutting are performed with conventional bur. Each patient will be given a questionnaire to fill out for each day starting from the day of surgery for 7 days postoperatively to assess the quality of life. They will be also requested to note down the details of analgesic intake. Hemorrhage control during surgery will be assesed. Clinical and radiographic examinations will be performed every 3, 6 and 12 months to evaluate any evidence of signs and/or symptoms and after 12 month follow up post operative CBCT taken to evaluate volume reduction of lesion postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with no general medical contra-indications for oral surgical procedures (ASA-1 or ASA-2).
2. Patients of age 16 years and above.
3. The tooth to be treated surgically should have a periradicular lesion of strictly endodontic origin (chronic apical periodontitis).
4. The nonsurgical re-treatment was judged unfeasible or had previously failed.
5. The tooth had an adequate final restoration with no clinical evidence of coronal leakage.
6. The apical area of the root canal should be devoid of the presence of a post for at least 6 mm.
7. Patients with no acute symptoms.

Exclusion Criteria:

1. Unrestorable tooth.
2. Fractured / perforated tooth.
3. Apicomarginal defects.
4. Through & through lesions.
5. Teeth with deep pockets.
6. Serious medical illness(uncontrolled/poorly controlled diabetes, unstable or life threatening conditions or requiring antibiotic prophylaxis).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment | Till 1 week after surgery
  By quality of life questionnaire(Igor Tsesis et al)
Postoperative healing | 12 months
  2D radiographic healing by Rud et al and Molven et al criteria and 3D healing by modified PENN 3D criteria

SECONDARY OUTCOMES:
hemorrhage control | during surgery
  assessed by scores used by Vy et al

CONTACTS AND LOCATIONS:
Overall Officials: JAYA BHARATHI, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES, ROHTAK
Locations (1):
- Post graduate institute of dental sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No